CLINICAL TRIAL: NCT06207409
Title: Program for Alleviating and Reducing Trauma, Stress, and Substance Use (PARTS-SUD)
Brief Title: Program for Alleviating and Reducing Trauma, Stress, and Substance Use
Acronym: (PARTS-SUD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Foundation for Self Leadership (Other)
Responsible Party: Principal Investigator, Zev Schuman Olivier, Director, Center for Mindfulness and Compassion, Cambridge Health Alliance
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHA-IRB-23-24-237
Record Dates: First submitted 2023-09-07; First posted 2024-01-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-01

CONDITIONS: PTSD; Substance Use Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PARTS-SUD Arm (Experimental): The Program for Alleviating and Reducing Trauma, Stress and Substance Use (PARTS-SUD) is a 12-week, Internal Family Systems-based, group intervention with 6 individual clinical sessions on a biweekly basis.
  Interventions: Behavioral: PARTS-SUD

INTERVENTIONS:
Behavioral: PARTS-SUD — The Program for Alleviating and Reducing Trauma, Stress and Substance Use (PARTS-SUD) is a 12-week, Internal Family Systems-based, group intervention with 6 individual clinical sessions on a biweekly basis.

SUMMARY:
This single-arm study will test the preliminary efficacy of a virtually delivered, live-online 12-week group model of Internal Family Systems (IFS) for individuals with posttraumatic stress disorder (PTSD) and substance use disorders (Program for Alleviating and Reducing Trauma, Stress, and Substance Use, PARTS-SUD).

Participants will be in a group for 12 weeks and will be asked to complete survey sessions at baseline and during week 4, 8 and 12.

DETAILED DESCRIPTION:
The investigators have conducted a single arm study of a 16 week PARTS group-based program for PTSD symptoms, which demonstrated large effect reductions on PTSD symptoms, disturbances in self-organization (DSO), disassociation, emotion dysregulation, suicide risk, anxiety, depression, and increases in decentering and self-compassion. A randomized control trial (RCT) of PARTS groups vs. a control is currently underway and will complete by September 2023. This will be a single-arm feasibility and acceptability pilot study of PARTS for PTSD among patients with substance use disorders.

While 16 weeks is the typical length for PTSD intervention trials, the average treatment length for PTSD-SUD population studies is only 12 weeks given higher risk of attrition with longer treatments for substance use disorder (SUD). Clinically, the group is anticipated to have the most impact on symptoms between weeks and 12 based on the curriculum and practices during those sessions, so the investigators will pilot a 12 week group in this study. Similar to past PARTS studies, participants will also have every other week 50 minute individual counseling sessions. Since IFS and group psychotherapy are established modalities and the pilot trial for PARTS established its evidence as a program with a clinically meaningful effect, this feasibility and acceptability study will primarily focus on the engagement and acceptability of the intervention among patients with PTSD-SUD. Both group and individual sessions will be billed to insurance as per standard Cambridge Health Alliance (CHA) outpatient clinical protocols. To reduce burden from past studies, the investigators will not conduct Clinician-Administered PTSD Scale (CAPS-5) interviews, but solely use self-report measures (PTSD Checklist For DSM-5, PCL-5 and Computerized Adaptive Testing for PTSD, CAT-PTSD), which have a high level of correlation with CAPS-5.

The investigators aim to have 10-12 participants allocated to start the program aiming for 70% of completion of the study intervention (defined as 75% completion of sessions) and 70% completion of week 12 assessments with adequate intervention acceptability. After participants have completed all baseline screenings, assessments and the informed consent procedure, a study staff member will contact them to begin the virtual program delivered in real time over the secure, HIPAA compliant video conference (e.g. Google Meets, Zoom).

Surveys, Procedures and Duration The duration of the study period is 12 weeks (see Figure 1). Participants will complete screening surveys and a long survey battery at baseline; survey batteries (approximately 62 minutes) at study Week 4, 8 and 12; and weekly substance use and craving self-report assessments.

All study procedures (screening, consent and assessments) can be conducted virtually, by videoconference and online through the secure REDCap survey database. These procedures may also be conducted in-person at a CHA community mental health center, and/or at the Center for Mindfulness and Compassion (CMC, 350 Commerce Place, Malden, MA).

ELIGIBILITY:
Inclusion Criteria:

* Able to bill insurance for group psychotherapy and individual psychotherapy at CHA;
* Currently or willing to become a patient of CHA primary care or behavioral health care (as defined by an active CHA EPIC EHR record);
* Have a current diagnosis of PTSD OR a CAT-MH PTSD>58;
* Have a current diagnosis of a substance use disorder (SUD), positive Alcohol Use Disorders Identification Test AUDIT-C item about 5 or more drinks at once OR positive toxicology for or self-report of illicit drugs in the past year, or current treatment with medications for OUD, including buprenorphine, naltrexone or methadone.
* Have sufficient English fluency and literacy skills to understand the consent process, procedures and questionnaires and have the ability to provide written informed consent;
* Have access to the internet and an electronic device with adequate data capacity; to complete questionnaires online and attend online video conference groups;
* Must be available and willing to attend 10 of 12 scheduled online group sessions for 12 weeks; and
* Must be available and willing to complete the online computerized assessments and phone interviews.

Exclusion Criteria:

* Inability to complete an informed consent assessment AND/OR inability to complete baseline study assessment procedures (due to cognitive deficit, non-proficiency in English literacy, or for any other reason);
* Current participation in another experimental research study;
* Expected medical hospitalization in the next four months from enrollment period;
* Expected incarceration in the next four months from enrollment period;
* Individuals who are pregnant with a due date within 16 weeks after study consent;
* Insufficient level of severity of PTSD symptoms: PTSD score of less than 33 on the PTSD Checklist for DSM-V (PCL-5) at screening visit will require clinical review to consider eligibility;
* Insufficiently stable housing or internet connection to join at least 10 sessions;
* Inability to participate safely in the study intervention and without disrupting the group (in the opinion of principal investigator OR meeting any of the following criteria):
* Past year history of a psychotic disorder or clinician confirmed active psychosis (Severe level of psychosis on PSY-S-CAT > 60 will require clinical assessment prior to participation in the program)
* Bipolar I disorder history or current severe level of mania on CAT-M/H (>70) will require of a clinical assessment prior to participation in the program
* Acute suicidality with intent will be excluded from the study (Columbia Suicide Rating Scale items 4-6 positive);
* Self-injurious behavior in past three months will require clinical assessment prior to participation in the program;
* Acute homicidality with plan and/or intent;
* Inpatient hospitalization for mental health, substance use, suicide attempt or self-harm within past three months;
* Severe Borderline Personality Disorder or other severe personality disorder with clinical history that would suggest potential disruptions within the group (would require clinical review);
* Inability to join a group without intoxication; and/or
* History of charges for perpetrating intimate partner violence will require clinical assessment prior to participation in the program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Completion Rate | 12 weeks
  The primary aim of this study is to examine the feasibility of a live-online version of the PARTS program defined as 70% of participants completing at least 75% (9/12) of groups.

SECONDARY OUTCOMES:
Assessment completion | 12 weeks
  Feasibility as measured by greater than or equal to 70% of participants completing post study assessments
Acceptability | 12 weeks
  Acceptability of the intervention as measured by a Theoretical Framework for Acceptability (TFA) overall acceptability item mean score > 3.5 out of 5.
Engagement | 12 weeks
  Satisfaction questionnaire with at least a mean of 7.5 out of 10 on being willing to recommend the program to a friend.

OTHER OUTCOMES:
PTSD symptom severity | 12 weeks
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure assessing symptom severity of PTSD. A total score of 31-33 or higher suggests that an individual may benefit from PTSD treatment.
Disassociation | 12 weeks
  The Multiscale Dissociation Inventory (MDI) is The MDI is a 30-item self-report test of dissociative symptomatology. The scale measures the following 5 aspects: Disengagement, Identity Dissociation, Emotional Constriction, Memory Disturbance, and Depersonalization/Derealization. A score of 15 or higher for the Identity Dissociation scale is suggestive of those with Dissociative Identity Disorder (DID). Each MDI symptom item is rated based on frequency of occurrence over the prior month, using a Likert scale ranging from 1 (never) to 5 (very often).
Disturbance in Self-Organization | 12 weeks
  The International Trauma Questionnaire (ITQ) is an 18-item self-report survey based on the criteria for Complex PTSD outlined in the International Classification of Diseases, 11th edition (ICD-11). This questionnaire is designed to differentiate between symptoms of PTSD and those of Complex PTSD. A diagnosis of PTSD can be determined if the respondent endorses questions related to symptoms of re-experiencing, avoidance, sense of current threat, or functional impairment. On the other hand, a diagnosis of Complex PTSD may be indicated if the respondent endorses questions pertaining to affective dysregulation, negative self-concept, disturbances in relationships, or disturbances in self-organization.
Addiction Severity | 12 weeks
  The Brief Addiction Monitor (BAM) is a self-report questionnaire consisting of 17 items that assess an individual's level of substance use, as well as the presence of risk and protective factors related to addiction. This scale provides scores in three domains: substance use, risk factors, and protective factors. In the substance use domain, scores range from 0 to 12, with higher scores indicating greater levels of substance use. For the risk factors domain, scores range from 0 to 24, with higher scores indicating a greater number of risk factors present. Conversely, in the protective factors domain, scores also range from 0 to 24, with higher scores indicating a greater number of protective factors present.

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Malden, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No